CLINICAL TRIAL: NCT01120418
Title: A Randomized, Contralateral Study To Evaluate Corneal Endothelial Cell Density Changes In Healthy Subjects, When Administered 0.6% ISV-403 Three Times Daily For Five Days
Brief Title: Corneal Endothelial Cell Density Changes In Healthy Subjects, When Administered ISV-403 for 5 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 507
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Endothelial cell density; screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Besifloxacin Ophthalmic Suspension 0.6% (Experimental): Topical ocular administration three times daily (TID) for 5 days
  Interventions: Drug: Besifloxacin Ophthalmic Suspension 0.6%

INTERVENTIONS:
Drug: Besifloxacin Ophthalmic Suspension 0.6% — administered 3 times a day for 5 days to one eye.
  Other Names: ISV-403

SUMMARY:
The objective of this study is to evaluate the effect on corneal endothelial cell density changes when ISV-403 is administered for five (5) days compared to no drug treatment, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have pin-holed Snellen visual acuity equal to or better than 20/40, in both eyes
* Must be in good health (no current or past relevant medical/ocular history) based on the judgment of the Investigator
* Must be willing to discontinue contact lens wear for the duration of the study

Exclusion Criteria:

* Known hypersensitivity to fourth generation fluoroquinolone (SS734) or to any of the ingredients in the study medication Investigator determines could interfere with the study
* History of extended or continuous wear contact lens use other than silicone hydrogels
* History of intraocular surgery
* Any topical ophthalmic medication, including tear substitutes, that cannot be discontinued during the study
* Participation in an ophthalmic drug or device research study within the 30 days prior to entry in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density change between treatment group. | Baseline, 5 days
  Difference in the change from baseline in endothelial cell density between eyes treated with besifloxacin ophthalmic suspension and untreated fellow eyes.

SECONDARY OUTCOMES:
Endothelial cell density change within treatment group | Baseline, 5 days
  Change from baseline in endothelial cell density within eyes treated with besifloxacin ophthalmic suspension and within untreated fellow eyes.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States